CLINICAL TRIAL: NCT04654234
Title: Total-body PET/CT Imaging Using the uEXPLORER in Non-small Cell Lung Cancer Patients Treated by Induction Chemotherapy Plus Nivolumab and Definitive Concurrent Chemoradiotherapy
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Clinical Professor, Sun Yat-sen University
Other Study IDs: GASTO-1067
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Total-body PET/CT; uEXPLORER; Nivolumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Total-body PET/CT (uExplorer): Patients with locally advanced NSCLC will receive total-body PET/CT (uExplorer) scans before, during and after the treatment
  Interventions: Device: Total body PET/CT (uExplorer)

INTERVENTIONS:
Device: Total body PET/CT (uExplorer) — A total-body positron emission tomography/computed tomography (PET/CT) scanner (uEXPLORER) with a 192-cm scan range was applied for cancer diagnosis, organ function assessment and treatment outcome prediction. The total-body PET scanner can acquire scans with lower administered activity or short acquisition time, total-body dynamic acquisition at a longer delayed time point, and high detectability of exiguous changes of the whole body, and tumor as well.

SUMMARY:
The prospective study aims to explore the value of total-body PET/CT dynamic imaging (uExplorer) in assessing tumor metabolic heterogeneity and predicting prognosis for patients with locally advanced, unresectable non-small cell lung cancer (stage III) treated by neoadjuvant chemotherapy plus nivolumab and definitive concurrent chemoradiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures;
* Patients aged 18~75 years old;
* had histologically or cytologically confirmed non-small cell lung cancer;
* Without prior chemotherapy, radiotherapy, surgery, targeted therapy or immunotherapy;
* Life expectancy ≥12 weeks;
* World Health Organization (WHO) Performance Status of 0 or 1;
* had unresectable stage III disease according to the 8th edition of the American Joint Committee on Cancer staging system;
* Women should be non-breast feeding during the study period;
* Women of reproductive age (WOCBP) must agree to comply with the contraceptive method during the study treatment and for a period of 5 months following the last administration of the study treatment;
* Men who have sex with WOCBP must agree to comply with the contraceptive method during the study treatment and for 7 months after the last administration of the study treatment;
* Absolute neutrophil count ≥1500/uL, hemoglobin ≥9.0mg/dL, platelet ≥100000/uL;
* Serum creatinine clearance >50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976);
* Serum bilirubin ≤1.5 x upper limit of normal (ULN), Aspartate Transaminase(AST) and Alanine Transaminase(ALT) ≤2.5 x ULN;
* Forced expiratory volume in 1 second (FEV1) ≥800ml;

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless it is an observational(non-interventional) clinical study;
* Mixed small cell and non-small cell lung cancer histology;
* Prior exposure to any anti-programmed cell death protein(PD)-1 or anti- PD-L1 antibody;
* Active or prior documented autoimmune disease within the past 2 years;
* Active or prior documented inflammatory bowel disease (eg. Crohn's disease, ulcerative colitis);
* History of primary immunodeficiency;
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses;
* History of another primary malignancy within 5 years, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study;
* Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control;
* Any situation not suitable for this study judged by researchers;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced non-small cell lung cancer patients treated by neoadjuvant chemotherapy plus nivolumab and definitive concurrent chemoradiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Patlak-Ki (Ki) | From enrollment to 1 year after radiotherapy
  The prognostic role of Patlak-Ki and its dynamic change during treatment

SECONDARY OUTCOMES:
standardized uptake value (SUV) | From enrollment to 1 year after radiotherapy
  The prognostic role of SUV and its dynamic change during treatment
metabolic tumor volume (MTV) | From enrollment to 1 year after radiotherapy
  The prognostic role of MTV and its dynamic change during treatment
total lesion glycolysis (TLG) | From enrollment to 1 year after radiotherapy
  The prognostic role of TLG and its dynamic change during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Le Chevalier T, Arriagada R, Quoix E, Ruffie P, Martin M, Tarayre M, Lacombe-Terrier MJ, Douillard JY, Laplanche A. Radiotherapy alone versus combined chemotherapy and radiotherapy in nonresectable non-small-cell lung cancer: first analysis of a randomized trial in 353 patients. J Natl Cancer Inst. 1991 Mar 20;83(6):417-23. doi: 10.1093/jnci/83.6.417. PMID 1847977
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Liao ZX, Komaki RR, Thames HD Jr, Liu HH, Tucker SL, Mohan R, Martel MK, Wei X, Yang K, Kim ES, Blumenschein G, Hong WK, Cox JD. Influence of technologic advances on outcomes in patients with unresectable, locally advanced non-small-cell lung cancer receiving concomitant chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):775-81. doi: 10.1016/j.ijrobp.2009.02.032. Epub 2009 Jun 8. PMID 19515503
- [Background] Zhang X, Xie Z, Berg E, Judenhofer MS, Liu W, Xu T, Ding Y, Lv Y, Dong Y, Deng Z, Tang S, Shi H, Hu P, Chen S, Bao J, Li H, Zhou J, Wang G, Cherry SR, Badawi RD, Qi J. Total-Body Dynamic Reconstruction and Parametric Imaging on the uEXPLORER. J Nucl Med. 2020 Feb;61(2):285-291. doi: 10.2967/jnumed.119.230565. Epub 2019 Jul 13. PMID 31302637
- [Background] Zhang YQ, Hu PC, Wu RZ, Gu YS, Chen SG, Yu HJ, Wang XQ, Song J, Shi HC. The image quality, lesion detectability, and acquisition time of 18F-FDG total-body PET/CT in oncological patients. Eur J Nucl Med Mol Imaging. 2020 Oct;47(11):2507-2515. doi: 10.1007/s00259-020-04823-w. Epub 2020 May 18. PMID 32424483
- [Background] Zhang X, Cherry SR, Xie Z, Shi H, Badawi RD, Qi J. Subsecond total-body imaging using ultrasensitive positron emission tomography. Proc Natl Acad Sci U S A. 2020 Feb 4;117(5):2265-2267. doi: 10.1073/pnas.1917379117. Epub 2020 Jan 21. PMID 31964808
- [Derived] Wang D, Mo Y, Liu F, Zheng S, Liu H, Li H, Guo J, Fan W, Qiu B, Zhang X, Liu H. Repeated dynamic [18F]FDG PET/CT imaging using a high-sensitivity PET/CT scanner for assessing non-small cell lung cancer patients undergoing induction immuno-chemotherapy followed by hypo-fractionated chemoradiotherapy and consolidative immunotherapy: report from a prospective observational study (GASTO-1067). Eur J Nucl Med Mol Imaging. 2024 Nov;51(13):4083-4098. doi: 10.1007/s00259-024-06819-2. Epub 2024 Jul 2. PMID 38953934